CLINICAL TRIAL: NCT03145597
Title: Survival Rate of Adhesively Luted Veneers, an In-vivo Study
Brief Title: Survival Rate of Adhesively Luted Veneers
Acronym: facings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Marco Gresnigt, dr., University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Laminate veneers
Record Dates: First submitted 2012-06-12; First posted 2017-05-09 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Tooth Fracture
Keywords: facings; veneers; laminates; existing; restorations; esthetics; dental
MeSH Terms: conditions — Tooth Fractures

STUDY DESIGN:
Intervention Model Description: split mouth comparison
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laminate veneer of composite (Experimental): Laminate veneer of composite (Estenia, Kuraray Dental), composite laminate veneer, 2-4-6 veneers per patient will be made.
  Interventions: Device: Laminate veneer of composite
- Laminate veneer of ceramic (Experimental): laminate of ceramic (Empress Esthetic, Ivoclar Vivadent), ceramic laminate veneer, 2-4-6 veneers per patient will be made.
  Interventions: Device: Laminate veneer of ceramic

INTERVENTIONS:
Device: Laminate veneer of composite — Composite laminate veneers, 2-4-6 veneers per patient
  Arms: Laminate veneer of composite
Device: Laminate veneer of ceramic — laminate of ceramic (Empress Esthetic, Ivoclar Vivadent), ceramic laminate veneer, 2-4-6 veneers per patient will be made.
  Arms: Laminate veneer of ceramic

SUMMARY:
The aims of this clinical study are:

To evaluate the clinical performance between indirect composite and ceramic laminate veneers:

Main interests are:

* colour stability of the restoration (digital measurement in follow up)
* failure mode of the restoration
* wear of the restoration and antagonist

Hypothesis:

* The colour stability of indirect composite restorations will not be different from the ceramic restorations.
* The indirect composite restorations will not be more prone to failure than the ceramic restorations.
* Antagonist wear and restorative material wear will be similar for both ceramic and composite.

Material and Methods The laminates will be fabricated according to a specified protocol. In order to avoid possible noticeable differences in case of distinct levels of possible discoloration, a modified split mouth design is employed where the central incisors and the symmetric other teeth receive the same type of restoration. Randomization is based on the paired teeth and it is performed using the flip of a coin for the choice of material. Evaluation will be performed at baseline and at follow-up visits annually up to 2 years.

DETAILED DESCRIPTION:
Patient recruitment: Patients will be recruited from the university clinic.

Intake: If the patient is included in the study following the inclusion and exclusion criteria, the patient will be evaluated using the evaluation form. All the data will be collected and impressions will be made. Using the impressions, a wax up will be made on stone models indicating the restorations to be fabricated. With a transparent mould, the situation will be duplicated in the mouth with spot etching and composite. By using this protocol minimal loss of tooth material is guaranteed.

Tooth Preparation: After prophylaxis, the teeth will be prepared in a controlled manner using special depth cutting laminate preparation burs (Intensive, Switzerland). The margins will extend to half the way to the inter-proximal contact area. The shape of the cervical margins will be maintained in chamfer form. The incisal edge will be prepared 1.5 mm to create an overlap to the palatinal region for the translucency area in the laminate veneers.

Conditioning the tooth surface: Rubberdam will be placed. The preparation surfaces will be etched with 35% phosphoric acid, rinsed thoroughly and dried followed by the application of primer and the bonding agent.

Conditioning the existing restorations: The existing composite restaurations will be conditioned using tribochemical silicacoating (CoJet, 30µm SiOx, 3M ESPE) in a Dentoprep (Ronvig, Denmark) intraoral sandblaster. Following this the restauration will be conditioned by silanisation.

Conditioning the composite veneers: The inner surfaces of the indirect composite laminates will rinsed with alcohol and thereafter conditioned using tribochemical silicacoating (CoJet, 30µm SiOx, 3M ESPE) using an (Ronvig, Denmark) intra-oral sandblaster. The sandblasting will be approx 13 sec until the inner surface of the restoration change colour visually. Following this the inner surface will be conditioned by silanisation.

Conditioning the ceramic veneers: The inner surfaces of the ceramic laminates will be conditioned with hydrofluoric acid 5% and rinsed in neutralizing agent, ultrasonically cleaned and then silanized.

After insertion, the excess composite will be removed using handinstruments and finishing burs under continuous water-cooling. Finally the margins will be polished using diamond polishing-paste with a rotating rubber cup. The interproximal surfaces will be finished with Sof-Lex polishing disks and strips.

Cementing the restorations: The cementation medium will be a dual-cure aesthetic adhesive cement Variolink veneer. All adhesive restorations will be cemented using ultrasonic insertion techniques. Cementation of the indirect restorations will be performed according to a protocol presented in appendix 2: "Clinical procedures".

ELIGIBILITY:
Inclusion Criteria:

1. The veneers will be placed on central incisors, lateral incisors, canines in the maxilla. Indications will involve replacing worn, discoloured composite restorations and existing veneers, or correcting discoloured, malformed and/or misaligned teeth.
2. An indication for closure of the open space (diastema)
3. No obvious untreated caries, dental health problems (regularly checked by a dentist).
4. No untreated periodontal disease (allowed are DPSI 1, 2, 3-)
5. Good or moderate oral hygiene (plaque score of less than 30% in anterior region before treatment).
6. Endodontic treatment with good outcome (root canal densely filled with gutta-percha 0.5-1.5 mm from apex) with only a restoration on palatinal side.
7. The patient agrees with the research protocol (signing of an agreement form, appendix 4)
8. 18 Year and older.

Exclusion Criteria:

1. Patients with only one tooth to restore, or two central incisors.
2. Considerable horizontal and/or vertical mobility of abutment teeth: tooth mobility index score 2 or 3.
3. Considerable periodontal disease without treatment (DPSI 3+ and 4)
4. Endodontic treatment with extensive loss of tooth tissue (more than 2/3 of crown is restored with restoration material).
5. Restoration of whole crown, more than 2/3 of coronal part of the teeth is restored.
6. Patients that still want to bleach their teeth or bleached teeth less than 3 weeks before the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
survival rate of laminate veneers | up to 24 months
  fracture of teeth

CONTACTS AND LOCATIONS:
Overall Officials: Marco Gresnigt, Phd, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blatz MB, Sadan A, Kern M. Resin-ceramic bonding: a review of the literature. J Prosthet Dent. 2003 Mar;89(3):268-74. doi: 10.1067/mpr.2003.50. PMID 12644802
- [Background] Blatz MB, Sadan A, Maltezos C, Blatz U, Mercante D, Burgess JO. In vitro durability of the resin bond to feldspathic ceramics. Am J Dent. 2004 Jun;17(3):169-72. PMID 15301212
- [Background] Brendeke J, Ozcan M. Effect of physicochemical aging conditions on the composite-composite repair bond strength. J Adhes Dent. 2007 Aug;9(4):399-406. PMID 17847643
- [Background] Brentel AS, Ozcan M, Valandro LF, Alarca LG, Amaral R, Bottino MA. Microtensile bond strength of a resin cement to feldpathic ceramic after different etching and silanization regimens in dry and aged conditions. Dent Mater. 2007 Nov;23(11):1323-31. doi: 10.1016/j.dental.2006.11.011. Epub 2006 Dec 26. PMID 17188745
- [Background] Busscher HJ, Rinastiti M, Siswomihardjo W, van der Mei HC. Biofilm formation on dental restorative and implant materials. J Dent Res. 2010 Jul;89(7):657-65. doi: 10.1177/0022034510368644. Epub 2010 May 6. PMID 20448246
- [Background] Ccahuana VZ, Ozcan M, Mesquita AM, Nishioka RS, Kimpara ET, Bottino MA. Surface degradation of glass ceramics after exposure to acidulated phosphate fluoride. J Appl Oral Sci. 2010 Mar-Apr;18(2):155-65. doi: 10.1590/s1678-77572010000200010. PMID 20485927
- [Background] Carlen A, Nikdel K, Wennerberg A, Holmberg K, Olsson J. Surface characteristics and in vitro biofilm formation on glass ionomer and composite resin. Biomaterials. 2001 Mar;22(5):481-7. doi: 10.1016/s0142-9612(00)00204-0. PMID 11214759
- [Background] Drummond JL. Degradation, fatigue, and failure of resin dental composite materials. J Dent Res. 2008 Aug;87(8):710-9. doi: 10.1177/154405910808700802. PMID 18650540
- [Background] Dumfahrt H, Schaffer H. Porcelain laminate veneers. A retrospective evaluation after 1 to 10 years of service: Part II--Clinical results. Int J Prosthodont. 2000 Jan-Feb;13(1):9-18. PMID 11203615
- [Background] Dunne SM, Millar BJ. A longitudinal study of the clinical performance of porcelain veneers. Br Dent J. 1993 Nov 6;175(9):317-21. doi: 10.1038/sj.bdj.4808314. PMID 8251248
- [Background] Ernest CP, Holzmeier M, Willershausen B. In vitro shear bond strength of self-etching adhesives in comparison to 4th and 5th generation adhesives. J Adhes Dent. 2004 Winter;6(4):293-9. PMID 15779314
- [Background] Ferracane JL, Berge HX, Condon JR. In vitro aging of dental composites in water--effect of degree of conversion, filler volume, and filler/matrix coupling. J Biomed Mater Res. 1998 Dec 5;42(3):465-72. doi: 10.1002/(sici)1097-4636(19981205)42:33.0.co;2-f. PMID 9788511
- [Background] Ferracane JL, Hopkin JK, Condon JR. Properties of heat-treated composites after aging in water. Dent Mater. 1995 Nov;11(6):354-8. doi: 10.1016/0109-5641(95)80034-4. PMID 8595835
- [Background] Fradeani M. Six-year follow-up with Empress veneers. Int J Periodontics Restorative Dent. 1998 Jun;18(3):216-25. PMID 9728104
- [Background] Fradeani M, Redemagni M, Corrado M. Porcelain laminate veneers: 6- to 12-year clinical evaluation--a retrospective study. Int J Periodontics Restorative Dent. 2005 Feb;25(1):9-17. PMID 15736774
- [Background] Friedman MJ. A 15-year review of porcelain veneer failure--a clinician's observations. Compend Contin Educ Dent. 1998 Jun;19(6):625-8, 630, 632 passim; quiz 638. PMID 9693518
- [Background] Fucio SB, Carvalho FG, Sobrinho LC, Sinhoreti MA, Puppin-Rontani RM. The influence of 30-day-old Streptococcus mutans biofilm on the surface of esthetic restorative materials--an in vitro study. J Dent. 2008 Oct;36(10):833-9. doi: 10.1016/j.jdent.2008.06.002. Epub 2008 Jul 14. PMID 18621456
- [Background] Fuzzi M, Zaccheroni Z, Vallania G. Scanning electron microscopy and profilometer evaluation of glazed and polished dental porcelain. Int J Prosthodont. 1996 Sep-Oct;9(5):452-8. PMID 9108746
- [Background] Gopferich A. Mechanisms of polymer degradation and erosion. Biomaterials. 1996 Jan;17(2):103-14. doi: 10.1016/0142-9612(96)85755-3. PMID 8624387
- [Background] Goracci C, Sadek FT, Monticelli F, Cardoso PE, Ferrari M. Microtensile bond strength of self-etching adhesives to enamel and dentin. J Adhes Dent. 2004 Winter;6(4):313-8. PMID 15779317
- [Background] Gresnigt M, Ozcan M, Muis M, Kalk W. Bonding of glass ceramic and indirect composite to non-aged and aged resin composite. J Adhes Dent. 2012 Feb;14(1):59-68. doi: 10.3290/j.jad.a21418. PMID 21594236
- [Background] Guess PC, Stappert CF. Midterm results of a 5-year prospective clinical investigation of extended ceramic veneers. Dent Mater. 2008 Jun;24(6):804-13. doi: 10.1016/j.dental.2007.09.009. Epub 2007 Nov 19. PMID 18006051
- [Background] Gurel G. Predictable, precise, and repeatable tooth preparation for porcelain laminate veneers. Pract Proced Aesthet Dent. 2003 Jan-Feb;15(1):17-24; quiz 26. PMID 12680057
- [Background] Karlsson S, Landahl I, Stegersjo G, Milleding P. A clinical evaluation of ceramic laminate veneers. Int J Prosthodont. 1992 Sep-Oct;5(5):447-51. PMID 1290574
- [Background] Kawai K, Urano M. Adherence of plaque components to different restorative materials. Oper Dent. 2001 Jul-Aug;26(4):396-400. PMID 11504440
- [Background] Kramer N, Kunzelmann KH, Taschner M, Mehl A, Garcia-Godoy F, Frankenberger R. Antagonist enamel wears more than ceramic inlays. J Dent Res. 2006 Dec;85(12):1097-100. doi: 10.1177/154405910608501206. PMID 17122161
- [Background] Lateef SS, Boateng S, Hartman TJ, Crot CA, Russell B, Hanley L. GRGDSP peptide-bound silicone membranes withstand mechanical flexing in vitro and display enhanced fibroblast adhesion. Biomaterials. 2002 Aug;23(15):3159-68. doi: 10.1016/s0142-9612(02)00062-5. PMID 12102187
- [Background] Leloup G, Holvoet PE, Bebelman S, Devaux J. Raman scattering determination of the depth of cure of light-activated composites: influence of different clinically relevant parameters. J Oral Rehabil. 2002 Jun;29(6):510-5. doi: 10.1046/j.1365-2842.2002.00889.x. PMID 12071917
- [Background] Magne P, Belser UC. Novel porcelain laminate preparation approach driven by a diagnostic mock-up. J Esthet Restor Dent. 2004;16(1):7-16; discussion 17-8. doi: 10.1111/j.1708-8240.2004.tb00444.x. PMID 15259539
- [Background] Meijering AC, Creugers NH, Roeters FJ, Mulder J. Survival of three types of veneer restorations in a clinical trial: a 2.5-year interim evaluation. J Dent. 1998 Sep;26(7):563-8. doi: 10.1016/s0300-5712(97)00032-8. PMID 9754744
- [Background] Oh WS, Delong R, Anusavice KJ. Factors affecting enamel and ceramic wear: a literature review. J Prosthet Dent. 2002 Apr;87(4):451-9. doi: 10.1067/mpr.2002.123851. PMID 12011863
- [Background] Oilo G. Biodegradation of dental composites/glass-ionomer cements. Adv Dent Res. 1992 Sep;6:50-4. doi: 10.1177/08959374920060011701. PMID 1292463
- [Background] Onisor I, Bouillaguet S, Krejci I. Influence of different surface treatments on marginal adaptation in enamel and dentin. J Adhes Dent. 2007 Jun;9(3):297-303. PMID 17655069
- [Background] Ozcan M, Alander P, Vallittu PK, Huysmans MC, Kalk W. Effect of three surface conditioning methods to improve bond strength of particulate filler resin composites. J Mater Sci Mater Med. 2005 Jan;16(1):21-7. doi: 10.1007/s10856-005-6442-4. PMID 15754140
- [Background] Ozcan M, Barbosa SH, Melo RM, Galhano GA, Bottino MA. Effect of surface conditioning methods on the microtensile bond strength of resin composite to composite after aging conditions. Dent Mater. 2007 Oct;23(10):1276-82. doi: 10.1016/j.dental.2006.11.007. Epub 2006 Dec 15. PMID 17174388
- [Background] Passos SP, Valandro LF, Amaral R, Ozcan M, Bottino MA, Kimpara ET. Does adhesive resin application contribute to resin bond durability on etched and silanized feldspathic ceramic? J Adhes Dent. 2008 Dec;10(6):455-60. PMID 19189676
- [Background] Peumans M, De Munck J, Fieuws S, Lambrechts P, Vanherle G, Van Meerbeek B. A prospective ten-year clinical trial of porcelain veneers. J Adhes Dent. 2004 Spring;6(1):65-76. PMID 15119590
- [Background] Rinastiti M, Ozcan M, Siswomihardjo W, Busscher HJ. Immediate repair bond strengths of microhybrid, nanohybrid and nanofilled composites after different surface treatments. J Dent. 2010 Jan;38(1):29-38. doi: 10.1016/j.jdent.2009.08.009. PMID 19735692
- [Background] Rinastiti M, Ozcan M, Siswomihardjo W, Busscher HJ, van der Mei HC. Effect of biofilm on the repair bond strengths of composites. J Dent Res. 2010 Dec;89(12):1476-81. doi: 10.1177/0022034510381395. Epub 2010 Oct 12. PMID 20940354
- [Background] Souza RO, Ozcan M, Michida SM, de Melo RM, Pavanelli CA, Bottino MA, Soares LE, Martin AA. Conversion degree of indirect resin composites and effect of thermocycling on their physical properties. J Prosthodont. 2010 Apr;19(3):218-25. doi: 10.1111/j.1532-849X.2009.00551.x. Epub 2009 Dec 21. PMID 20040031
- [Background] Takeshige F, Kawakami Y, Hayashi M, Ebisu S. Fatigue behavior of resin composites in aqueous environments. Dent Mater. 2007 Jul;23(7):893-9. doi: 10.1016/j.dental.2006.06.031. Epub 2006 Sep 27. PMID 17007919
- [Background] Wakiaga J, Brunton P, Silikas N, Glenny AM. Direct versus indirect veneer restorations for intrinsic dental stains. Cochrane Database Syst Rev. 2004;(1):CD004347. doi: 10.1002/14651858.CD004347.pub2. PMID 14974066
- [Background] Walls AW, Murray JJ, McCabe JF. Composite laminate veneers: a clinical study. J Oral Rehabil. 1988 Sep;15(5):439-54. doi: 10.1111/j.1365-2842.1988.tb00180.x. PMID 3244054